CLINICAL TRIAL: NCT03827824
Title: Intervention Study to Measure the Effect on Perception of Pain and Anxiety in Women With Indication for Diagnostic Hysteroscopy Through the Use of Virtual Reality
Brief Title: Virtual Reality on Perception of Pain and Anxiety by Hysteroscopy
Acronym: Hysteroscopy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Complete collection of study patients
Sponsor: Universidad Francisco de Vitoria (Other)
Collaborators: Jesús Pelazas Hernández (Unknown); David Varillas Delgado (Unknown); Ignacio Cristóbal García (Unknown); Teresa González Casado (Unknown); Ignacio Cristóbal Quevedo (Unknown); Agustina Alonso Bermejo (Unknown); Marina Ronchas Martínez (Unknown)
Responsible Party: Principal Investigator, David Varillas Delgado, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12.18
Record Dates: First submitted 2019-01-24; First posted 2019-02-01 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2022-07

CONDITIONS: Uterine Diseases
Keywords: Virtual Reality; Hysteroscopy; Pain; Anxiety
MeSH Terms: conditions — Uterine Diseases; Pain; Anxiety Disorders | interventions — Hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hysteroscopy & Virtual reality glasses (Experimental): Hysteroscopy with use of virtual reality glasses
  Interventions: Device: Hysteroscopy & virtual reality glasses; Device: Hysteroscopy
- Hysteroscopy (Active Comparator): Hysteroscopy without use of virtual reality glasses
  Interventions: Device: Hysteroscopy

INTERVENTIONS:
Device: Hysteroscopy & virtual reality glasses — Hysteroscopy. Virtual reality glasses. VAS. STAI scale.
  Arms: Hysteroscopy & Virtual reality glasses
Device: Hysteroscopy — Hysteroscopy. VAS. STAI scale.

SUMMARY:
Randomized intervention trial with a calculated sample size of 90 women aged between 18 and 75 years and medical criteria for performing a diagnostic hysteroscopy according to the Gynecology and Obstetrics Spanish Society (SEGO).

Nowadays the investigators known that acute pain requires cognitive attention for its perception, a patient's state of anxiety depends on the subjective capacity to cope with the process and that environments created with virtual reality can cause a cognitive distraction that diminishes the perception of pain as well as a subjective psychological illusion that diminishes the anxiety that motivates the procedure.

For all the above, the investigators will study as a main objective the differences between the use of virtual reality through the use of virtual reality glasses "Oculus go model", to reduce the perception of pain and anxiety motivated by the performance of a outpatient hysteroscopy versus clinical practice. It is usual not to use analgesia, using the VAS pain scale and the STAI (State-Trait Anxiety Inventory) questionnaire to assess the state of anxiety before and after the test. In addition, as secondary objectives, the investigators will compare different aspects such as surgical time used, determination of vital signs, satisfaction studies ...

DETAILED DESCRIPTION:
A Cochrane review (included 32 clinical trials and 3304 patients) concluded that there was no effective and safe treatment for pain relief in patients undergoing outpatient hysteroscopy. In the same way, The Gynecology and Obstetrics Spanish Society (SEGO) discourages the routine use of analgesics prior to the test or the use of local anesthesia or sedation, since neither improves the pain nor the satisfaction of the patients in this type of test.

Nowadays, is knowed that acute pain requires cognitive attention for its perception, a patient's state of anxiety depends on the subjective capacity to cope with the process and that environments created with virtual reality can cause a cognitive distraction that diminishes the perception of pain as well as a subjective psychological illusion that diminishes the anxiety that motivates the procedure.

With all this, the investigators intend to assess through this study if patients with medical indication for diagnostic hysteroscopy can benefit from the use of Virtual Reality for the decrease in their perception of pain, anxiety or increase in the degree of satisfaction with their performance.

1. - Design: Randomized intervention clinical trial
2. - Sample: by contrast of hypothesis, a sample size of 90 women with an established medical indication for outpatient hysteroscopy was determined. They were randomized using excel software. As criteria of inclusion, those of SEGO with ages between 18 and 75 years were used. Criteria of exclusion those of the test, presenting some type of illness or disability that contraindicate the use of Virtual Reality (blindness, deafness, epilepsy, etc), voluntary wish of no inclusion or inability to understand the study.
3. - Methodology:

   * parameters to analyze:

     * the average decrease in the perception of pain in both groups using the Visual Analogue Scale (VAS) with determinations at the end, at 15 and 30 minutes.
     * the average decrease in the perception of the state of anxiety using the State-Trait Anxiety Inventory (STAI) questionnaire prior to the performance of the test and after it.
     * Modifications in the degree of satisfaction with the test by means of a STAI questionnaire included in the protocol of the Gynecology Service of El Escorial University Hospital.
     * Changes in parameters such as blood pressure, heart rate and oxygen saturation before, during and after hysteroscopy.
     * The influence of different circumstances such as age, parity, on the painful perception, state of anxiety or degree of satisfaction in both arms of the study.
   * A 5 mm Bettocchi hysteroscope model will be used as a physiological serum distension medium and initial irrigation pressures of 75 mm Hg.
   * Semi-rigid 5 Charr instruments (scissors, grasping forceps and biopsy).
   * Oculus Go virtual reality glasses.
   * The recruitment time will be that necessary to obtain the sample size.
   * The patients will be given the STAI anxiety scale that will be completed prior to accessing the room. Once sitting on the examination table, a pulse oximeter will be placed on the left index finger, a cuff for measuring blood pressure on the right arm, and in the selected group virtual reality glasses, the first determination of blood pressure, heart rate and oxygen saturation is made at this time and will be repeated when accessing the endometrial cavity and immediately after removing the hysteroscope. After completing the test, still sitting and removed the virtual reality components will be given VAS for pain determination during the test. After dressing, the pain will be assessed using VAS at 15 and 30 minutes after the end of the test. Before leaving, a new STAI anxiety state will be delivered that will complete as well as respond to the two questions of the satisfaction protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women with an established indication for diagnostic hysteroscopy according to the Spanish Society of Gynecology and Obstetrics (SEGO) criteria collected in its document of consensus, updated in 2013, with the title of "Hysteroscopy in consultation".
* Age between 18 and 75 years.
* Suitable cultural level for the understanding of the characteristics of the study.
* Signature of informed consent.

Exclusion Criteria:

* Not be within the criteria established by SEGO for the realization of a hysteroscopy diagnostic.
* Existence of contraindication for hysteroscopy.
* Present some type of disease or disability that can intervene in the object of the study: visual deficit, auditory or sensory severe, illnesses or mental syndromes.
* Having suffered seizures, loss of knowledge, or other symptoms related to epileptic disorders that discourages the use of virtual reality glasses.
* Women who cannot tolerate the pain at the beginning and during hysteroscopy.
* Not signature of informed consent.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-03-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline VAS at 30 minutes.
  Visual Analogue Scale: A measurement instrument that tries to measure a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured.This scale is between the values 0 to 10, being 0 the greatest pain possible and 10 the least pain. It is categorized into several sections, being intense pain 0-3, moderate pain 4-7 and low pain 8-10.
State-Trait Anxiety Inventory (STAI) | Change from baseline STAI scale at 30 minutes.
  State-Trait Anxiety Inventory (STAI): A psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Scores range from 20 to 80, with higher scores correlating with greater anxiety. Each measure has a different rating scale. The 4-point scale for S-anxiety is as follows: 1.) not at all, 2.) somewhat, 3.) moderately so, 4.) very much so. The 4-point scale for T-anxiety is as follows: 1.) almost never, 2.) sometimes, 3.) often, 4.) almost always.

SECONDARY OUTCOMES:
Systolic and Diastolic blood pressure | Changes of systolic and diastolic blood pressure from baseline at 30 minutes.
  Analize both blood pressures (systolic and diastolic) modifications in patients of study, experimental and active comparator groups.
Cardiac frequency | Changes of cardiac frequency from baseline at 30 minutes.
  Analize cardiac frenquence modifications in intervention group previous procedure, during the procedure and at the end of procedure.
Oxygen saturation | Changes of oxygen saturation from baseline at 30 minutes.
  Analize oxygen saturation modifications in intervention group previous procedure, during the procedure and at the end of procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Jesús V Pelazas Hernández, MD, Principal Investigator — Hospital El Escorial
Locations (1):
- David Varillas Delgado, Pozuelo de Alarcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided